CLINICAL TRIAL: NCT01400477
Title: Nicotinic Receptors and Schizophrenia: Phase II
Brief Title: Nicotinic Receptors and Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-0459; 5P50MH086383-02 (NIH); R01MH061412-05 (NIH); VA Merit Review grant (Other Grant/Funding Number: VA Merit Review grant)
Record Dates: First submitted 2011-07-14; First posted 2011-07-22 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Drug Trial; Smoking; Smoking Cessation; Cognition; Mental Focus
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Smoking; Smoking Cessation | interventions — 3-(2,4-dimethoxybenzylidene)anabaseine

STUDY DESIGN:
Intervention Model Description: Random allocation to a treatment and placebo group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The pharmacist places the treatment or placebo into identical coded vials. Only the pharmacist and the statistician have the code to identify of the treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DMXB-A-SR (Experimental): Study Drug: 3-2, 4 dimethoxybenzylidene anabaseine sustained release (DMXB-A-SR), 3-2, 4 dimethoxybenzylidene anabaseine sustained release (GTS-21)
  Interventions: Drug: DMXB-A-SR
- Arm #2: Placebo Comparator (Placebo Comparator): Inert capsule to resemble active drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DMXB-A-SR — Experimental Study Drug: 3-2, 4 dimethoxybenzylidene anabaseine sustained release (DMXB-A-SR)
  Other Names: GTS-21
  Arms: DMXB-A-SR
Other: Placebo — Placebo Comparator
  Arms: Arm #2: Placebo Comparator

SUMMARY:
The investigators hypothesize that sustained-release DMXB-A-SR (3-2,4 dimethoxybenzylidene anabaseine sustained release) will provide clinical improvement in cognition in patients with schizophrenia who are smokers and who are non-smokers. The study drug may also maintain abstinence from cigarette smoking and improve other symptoms in patients with schizophrenia.

DETAILED DESCRIPTION:
Patients with schizophrenia will be screened then enrolled for one week placebo trial in addition to their existing antipsychotic medication. If pill compliance is greater than 80%, then they will receive baseline clinical, cognitive, and brain imaging and all clinical laboratory examinations and a physical examination, vital signs, and cardiogram. Then patients will receive in a randomized double blind trial either DMXB-A-SR (3-2,4 dimethoxybenzylidene anabaseine sustained release) or placebo comparator in addition to their existing antipsychotic medication. After one month patients will receive repeat clinical, cognitive, and brain imaging testing and all clinical laboratory examinations and a physical examination, vital signs, and cardiogram.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be selected to be 18 to 65 years old and in good general health.
* Subjects who fulfill Diagnostic and Statistical Manual -IV-Text Revision (DSM-IV-TR) criteria for schizophrenia or schizoaffective disorder.
* Smokers will smoke at least 20 cigarettes per day.
* Non-smokers will also be enrolled.
* Subjects will have normal:

  * vital signs,
  * hematology,
  * serum chemistries,
  * EKG, and
  * urinalysis with a negative drug screen before entry into the study.
* Subjects will be fluent in English.
* Smoking subjects will be interested in stopping smoking in the near future and not interested in nicotine replacement therapy.

Exclusion Criteria:

* Subjects with histories of:

  * neurological illness,
  * liver disease,
  * severe hypertension (cut-off blood pressure 160/100) or
  * cardiac disease, or
  * renal failure (cut-off creatinine above 1.4).
* Subjects who currently meet DSM-IV-TR criteria for substance dependence other than nicotine, cannabis, or alcohol will be excluded.
* Women who are capable of pregnancy and not on acceptable forms of birth control will be excluded.
* Subjects being treated with Clozapine will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - UColorado Denver, Aurora, Colorado
  - University of Colorado-Anschutz Medical Campus, Department of Psychiatry, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: Yes
Individual patient description can be obtained from Robert.Freedman@ucdenver.edu. It will be available December 1, 2017.

REFERENCES:
- [Background] Olincy A, Harris JG, Johnson LL, Pender V, Kongs S, Allensworth D, Ellis J, Zerbe GO, Leonard S, Stevens KE, Stevens JO, Martin L, Adler LE, Soti F, Kem WR, Freedman R. Proof-of-concept trial of an alpha7 nicotinic agonist in schizophrenia. Arch Gen Psychiatry. 2006 Jun;63(6):630-8. doi: 10.1001/archpsyc.63.6.630. PMID 16754836
- [Background] Freedman R, Olincy A, Buchanan RW, Harris JG, Gold JM, Johnson L, Allensworth D, Guzman-Bonilla A, Clement B, Ball MP, Kutnick J, Pender V, Martin LF, Stevens KE, Wagner BD, Zerbe GO, Soti F, Kem WR. Initial phase 2 trial of a nicotinic agonist in schizophrenia. Am J Psychiatry. 2008 Aug;165(8):1040-7. doi: 10.1176/appi.ajp.2008.07071135. Epub 2008 Apr 1. PMID 18381905
- [Derived] Kem WR, Olincy A, Johnson L, Harris J, Wagner BD, Buchanan RW, Christians U, Freedman R. Pharmacokinetic Limitations on Effects of an Alpha7-Nicotinic Receptor Agonist in Schizophrenia: Randomized Trial with an Extended-Release Formulation. Neuropsychopharmacology. 2018 Feb;43(3):583-589. doi: 10.1038/npp.2017.182. Epub 2017 Aug 21. PMID 28825423

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DMXB-A-SR | Arm #2: Placebo Comparator
Started | 40 | 40
Completed | 38 | 40
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DMXB-A-SR | Arm #2: Placebo Comparator | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (12.4) | 43.2 (13.6) | 44.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 12 | 20
  Male | 32 | 28 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 10 | 16
  White | 32 | 30 | 62
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Neurocognitive Efficacy
Description: MATRICS CCB Neurocognitive T-score (Measurement and Treatment Research to Improve Cognition in Schizophrenia Consensus Cognitive Battery Statistically Adjusted-score). Higher scores indicate better neurocognitive functionality.
Time Frame: 4 weeks
Population: participants
Measure: Mean (Standard Deviation); unit: MATRICS Neurocognitive T score
Arm/Group | DMXB-A-SR | Arm #2: Placebo Comparator
Number analyzed (Participants) | 38 | 40
MATRICS Neurocognitive T score | 0.6 (5.8) | 2.1 (8.2)
Statistical Analysis 1: Comparison: DMXB-A-SR; Test type: Superiority; p = 0.89, ANOVA — A priori vape was <0.05; df 1, 37

2. Secondary Outcome: Inhibition of Auditory Evoked Potential P50 to Repeated Stimuli
Description: The P50 evoked response paired of auditory stimuli S1, S2, is measured. The inhibition is expressed as the ratio P50 S2 amplitude divided by P50 S1 amplitude.
Time Frame: 4 weeks
Population: Participants
Measure: Mean (Standard Deviation); unit: percentage of amplitude
Arm/Group | DMXB-A-SR | Arm #2: Placebo Comparator
Number analyzed (Participants) | 38 | 40
percentage of amplitude | 0.57 (0.12) | 0.52 (0.14)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Side Effects Questionnaire, complete blood count, urinalysis, and blood chemistry panel at 4 weeks
Arm/Group | DMXB-A-SR | Arm #2: Placebo Comparator
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes